CLINICAL TRIAL: NCT06846424
Title: A Clinical Study to Evaluate the Safety and Tolerability of SCT-001 CAR-T Cells in Patients with Recurrent and Refractory Epithelial Ovarian Cancer, Fallopian Tube Cancer, and Peritoneal Cancer.
Brief Title: SCT-001 CAR T Cells Therapy for Relapsed and Refractory Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Responsible Party: Principal Investigator, Rongyu Zang, MD,PhD, Doctor, Shanghai Gynecologic Oncology Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT-001 CAR-T OC
Record Dates: First submitted 2025-02-17; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Carcinoma; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCT-001 CAR-T intraperitoneal route of administration (Experimental): Patients receive SCT-001CAR-T cells via IP administration with or without lymphodepletion.
  Interventions: Biological: SCT-001 CAR-T cells
- SCT-001 CAR-T intravenous route of administration (Experimental): Patients receive SCT-001CAR-T cells via IV administration with or without lymphodepletion.
  Interventions: Biological: SCT-001 CAR-T cells

INTERVENTIONS:
Biological: SCT-001 CAR-T cells — SCT-001 CAR-T cells are autologous-derived CAR-T cell products, which transduce second-generation CAR targeting TAG-72 into patient autologous T cells by lentiviral transfection, and knock out immunosuppressive related genes by CRISPR/Cas9 technology to enhance the anti-tumor function of CAR-T cells.

SUMMARY:
This study is an open-label, dose-escalation, investigator-initiated phase I interventional clinical study. To evaluate the safety, tolerability and preliminary efficacy of SCT-001 CAR-T cell injection in subjects with relapsed and refractory epithelial ovarian, fallopian tube and peritoneal cancer, and to explore the pharmacokinetic characteristics, biomarker changes and immunogenicity of SCT-001 CAR-T cell injection in subjects with relapsed and refractory epithelial ovarian, fallopian tube and peritoneal cancer.

In this study, two trial cohorts were set up, cohort 1 was the intraperitoneal route of administration, and the subjects enrolled in cohort 1 needed to meet the conditions for intraperitoneal administration ((1) the subject had a large amount of ascites, (2) the subject was suitable for peritoneal catheterization, (3) the subject had no severe abdominal adhesions, and (4) the subject agreed to undergo intraperitoneal surgical catheterization for intraperitoneal administration); Cohort 2 is the intravenous route.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria for admission to this study:

Age≥ 18 years old;

* ECOG performance status score: 0~2 points or KPS score≥70 points;
* Relapsed or refractory epithelial ovarian, fallopian tube and peritoneal cancer confirmed by histology or cytology and have failed, are intolerant or have no standard treatment after standard therapy;
* Tumor tissue specimens or tumor samples can be obtained by tumor biopsy and other methods;
* Immunohistochemistry (IHC) staining confirmed that the tumor cells had positive TAG-72 expression (positive definition: >). IHC staining intensity of 1% tumor cells ≥2+);
* Estimated survival time of more than 3 months;
* At least one evaluable tumor lesion according to RECIST 1.1;
* Prior to treatment, major organ function met the following criteria (no blood transfusion, long-acting EPO, long-acting G-CSF therapy within 14 days prior to study drug administration, in the case of short-acting EPO, short-acting G-CSF, this criterion can be shortened to 7 days):
* complete blood count: Absolute neutrophil count (ANC) ≥1.5×109/L,, Absolute lymphocyte count (ALC) ≥ 0.5×109/L; hemoglobin (HGB) ≥ 80 g/L; Platelets (PLT) ≥ 75×109/L;
* Renal: serum creatinine ≤1.5× upper limit of normal range (ULN);
* Liver: total bilirubin ≤ 1.5× ULN (including patients with liver metastases or liver cancer), AST and ALT ≤ 2.5× ULN (liver metastases ≤5×ULN);
* Coagulation: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5× ULN, partially activated thromboplastin time (APTT) ≤ 1.5× ULN;
* Must be using adequate contraception during the study and for 6 months after the end of the study, have a negative serum pregnancy test within 7 days prior to proposed enrollment in the study, and must be a non-lactating subject.

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be admitted to this study:
* Those who are allergic to any component of SCT-001 CAR-T cell injection;
* Received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc., or participated in other clinical trials and received 5 half-lives of therapeutic drugs within 4 weeks prior to the first use of the study drug (4 weeks or 5 half-lives, whichever is shorter);
* Received treatment with traditional Chinese medicine or modern Chinese medicine preparations with anti-tumor indications in the label within 14 days before the first dose;
* The adverse reactions of previous anti-tumor therapy have not recovered to NCI CTCAE v5.0 grade evaluation ≤ grade 1 (except for toxicity that the investigator judges has no safety risk such as alopecia);
* Surgical procedure within 4 weeks prior to treatment or has not fully recovered from any previous invasive procedure;
* Central nervous system metastases or meningeal metastases with clinical symptoms, or other evidence that the subject's central nervous system metastases or meningeal metastases have not been controlled, and are judged by the investigator to be unsuitable for enrollment;
* Those with active infection (NCI CTCAE v5.0≥ grade 2) or any other person with suspected risk of infection as assessed by the investigator;
* Has a history of autoimmune disease, immunodeficiency, including a positive HIV test, or has other acquired, congenital immunodeficiency diseases, or has a history of organ transplantation;
* Subjects with active hepatitis B or active hepatitis C;
* Those who have used immune cell therapy in the past;
* History of severe cardiovascular disease, such as severe cardiac rhythm or conduction abnormalities (ventricular arrhythmia requiring clinical intervention, II.~III. degree atrioventricular block, etc.), myocardial infarction, history of coronary artery bypass surgery, heart failure, New York College of Cardiology (NYHA) grade II or above, left ventricular ejection fraction (LVEF) ≤50% and thrombosis found, male QTcF >450msec or female QTcF >470msec, etc.;
* Subjects with a history of severe cerebrovascular diseases such as stroke;
* Need to combine with other anti-tumor therapies (including various radiotherapy, chemotherapy, immunotherapy, targeted therapy, traditional Chinese medicine therapy, etc.);
* Previous clear history of neurological or psychiatric disorders, including epilepsy or dementia;
* In the opinion of the investigator, the subject has other reasons that make it unsuitable to participate in this clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 28 days
  The incidence of of DLT event, which is defined as toxic events related to SCT-001 CAR-T cell injection that occur within the DLT observation period (28 days after CAR-T cell injection), including general adverse events graded according to NCI CTCAE v5.0, cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS).
Incidence of adverse events | 24 months
  Toxicity within 24 months after CAR-T cell injection will be graded according to the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Change of CAR Copies | 12 months
  CAR Copies measured by qPCR (12 months after CAR-T infusion)
Objective response rate | 12 months
  The proportion of patients with complete response (CR) and partial response (PR) assessed by the investigator in accordance with the RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China